CLINICAL TRIAL: NCT05486455
Title: Evaluation of Lung Cancer CT Screening Performance Among Former and Current Smokers: a "Real Life" Study
Brief Title: Evaluation of Lung Cancer CT Screening Performance Among Former and Current Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DEPITAB
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT scan (Experimental)
  Interventions: Diagnostic Test: Low-dose chest CT scan

INTERVENTIONS:
Diagnostic Test: Low-dose chest CT scan — baseline, 1-year, 3-year and 5-year low-dose CT scan

SUMMARY:
Diagnostic performance of low-dose chest CT scan combined with lung-RADS classification (version 1.1) for lung cancer screening among former and current smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 50-80 years old
* Active smoker (≥ 15 PA) or former smoker (≥ 15 PA)

Exclusion Criteria:

* Recent history of chest CT scan (within 12 months)
* Person unable to climb 2 floors
* Weight > 140kg
* Personal history of cancer < 5 years (currently being monitored by thoracic imaging)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) | 5 years

SECONDARY OUTCOMES:
Sensitivity | 5 years
Specificity | 5 years
Early stage lung cancer detection rate (stage I and II) | 5 years
5-year survival rate of patients who have undergone thoracic surgery | 5 years
Rate of smoking-related co-morbidities detected on low-dose CT scan | 5 years
  smoking-related co-morbities = pulmonary emphysema, interstitial lung disease, atheromatous disease, hepatic steatosis and ascending aortic aneurysm.
Rate of additional examinations (including invasive diagnostic tests and surgery with benign results) | 5 years
Risk ratio of lung cancer | 5 years
Number of false positive results | 5 years
Penetration rate | 5 years
  number of subjects included / number of includible subjects
Smoking cessation rates | 5 years
EORTC QLQ-C30 score (version 3) | 5 years
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions.
  The EORTC QLQ-C30 is composed of 9 multi-item scales: 5 functioning scales (physical, role, cognitive, emotional and social), a global QOL scale, and 3 symptom scales (fatigue, pain and nausea/vomiting). In addition, several single item symptom measures are used.
  For the five functioning scales and the global quality of life scale, a higher score represents a better level of functioning. For the symptom scales and items, a high score corresponds to a higher level of symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Boyer, MD, Principal Investigator — Hopital Saint Joseph Marseille; Illies Bouabdallah, MD, Study Director — Hopital Saint Joseph Marseille
Locations (1):
- Hôpital Saint Joseph, Marseille, France